CLINICAL TRIAL: NCT00664703
Title: A Double-Blind, Double-Dummy, Placebo-Controlled, Dose Ranging Study of 7.5, 15, and 30 mg of Sublingual Lobeline in Adult ADHD Patients
Brief Title: Effectiveness of Lobeline in Treating Symptoms of ADHD in Adult Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yaupon Therapeutics (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: R43MH081553 (NIH); R43MH081553 (NIH); DATR BT-BU; 2007LOBADHD-201-US (Other: Yaupon Therapeutics, Inc.); 7-0432-F2L (Other: University of Kentucky Medical IRB)
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Dopamine Uptake Inhibitors; Dopamine; Methylphenidate; Mental Disorders Diagnosed in Childhood; Neurologic Manifestations; Attention Deficit and Disruptive Behavior Disorders; Hyperkinesis; Dyskinesias
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Neurodevelopmental Disorders; Neurologic Manifestations; Attention Deficit and Disruptive Behavior Disorders; Hyperkinesis; Dyskinesias | interventions — Lobeline; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Lobeline 7.5 mg (Experimental): Sublingual tablet
  Interventions: Drug: Lobeline sulfate
- Lobeline 15 mg (Experimental): Sublingual tablet
  Interventions: Drug: Lobeline sulfate
- Lobeline 30 mg (Experimental): Sublingual tablet
  Interventions: Drug: Lobeline sulfate
- Methylphenidate HCl 15 mg (Active Comparator): Capsule
  Interventions: Drug: Methylphenidate HCl
- Methylphenidate HCl 30 mg (Active Comparator): Capsule
  Interventions: Drug: Methylphenidate HCl
- Lobeline 0 mg (placebo) (Placebo Comparator): Sublingual tablet
  Interventions: Drug: Placebo
- Methylphenidate HCl 0 mg (placebo) (Placebo Comparator): Capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lobeline sulfate — Each laboratory day, participants will receive one capsule containing either methylphenidate HCl (15 or 30 mg) or placebo, and one sublingual tablet containing either lobeline (7.5, 15, or 30 mg) or placebo.
  Arms: Lobeline 15 mg; Lobeline 30 mg; Lobeline 7.5 mg
Drug: Methylphenidate HCl — Each laboratory day, participants will receive one capsule containing either methylphenidate HCl (15 or 30 mg) or placebo, and one sublingual tablet containing either lobeline (7.5, 15, or 30 mg) or placebo.
  Arms: Methylphenidate HCl 15 mg; Methylphenidate HCl 30 mg
Drug: Placebo — Each laboratory day, participants will receive one capsule containing either methylphenidate HCl (15 or 30 mg) or placebo, and one sublingual tablet containing either lobeline (7.5, 15, or 30 mg) or placebo.
  Arms: Lobeline 0 mg (placebo); Methylphenidate HCl 0 mg (placebo)

SUMMARY:
The study will evaluate the effectiveness of the nonstimulant medication lobeline in improving symptoms of attention deficit hyperactivity disorder in adults.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) affects approximately 8 million adults in the United States. Adults with ADHD may experience difficulty concentrating, poor organization ability, mood swings, and trouble completing work. If not managed properly, ADHD can lead to behavioral, emotional, academic, social, and work-related problems. Neurobiological research has shown that people with ADHD exhibit low levels of dopamine, a neurotransmitter of the brain that controls a person's ability to concentrate and focus on surroundings. Lobeline, a nonstimulant medication that acts to alter dopamine uptake, may be effective in improving abnormalities in brain dopamine levels. Although lobeline has been successfully used as a smoking cessation aid because of its ability to inhibit nicotine-induced hyperactivity, the effectiveness of lobeline as a treatment for ADHD has not been explored. This study will evaluate the effectiveness of lobeline in improving adult ADHD symptoms, specifically inattention, impulsivity, and memory problems. This study will also evaluate any side effects of lobeline treatment.

Participation in this study will last between 4 and 5 weeks, during which participants will attend 10 study visits at the General Clinical Research Center (GCRC). Participants will first undergo a medical evaluation visit that will include a physical exam, electrocardiogram (EKG), blood draw, urine testing, and breath sampling. Participants will then return for an orientation visit to complete questionnaires and to receive training on the computer and on memory tasks to be performed during later visits.

The next 7 visits will comprise the laboratory testing and medication treatment portion of the study. Each visit will last 4.5 hours and will include urine and breath sampling, computer and memory tasks, questionnaires, vital sign measurements, and medication distribution. Participants will be randomly assigned to take two different pills at each lab visit. One pill will be a placebo of lobeline or methylphenidate, a medication stimulant used in treating ADHD, and the other pill will be active lobeline or methylphenidate. Drug combinations and doses will vary each day, but participants will never receive two active pills on the same day. All participants will undergo a follow-up evaluation between 7 and 14 days after the final lab visit. The evaluation will include questions about side effects from study medication, breath and urine sampling, a blood draw, and a physical exam.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADHD, including degree of symptomatology, as determined by a structured clinical assessment based on the DSM-IV (SCID-1); supplemented by administration of the Schedule for Affective Disorders and Schizophrenia for School-Age Children, Epidemiologic version (KSADS-E) and administration of the Conners' Adult ADHD Rating Scale (CAARS);
* Healthy males or females aged 21 to 45 years;
* A body mass index (BMI) between 18 and 30;
* Ability and willingness to provide written consent, comply with study instructions, and commit to all study visits and procedures;
* Adequate means of contacting the investigator in case of emergency or have means to be contacted readily by the investigator;
* No medical contraindications determined by the following: an adequate medical history, a physical examination including vital signs, 12-lead electrocardiogram (ECG); complete blood count with differential liver function and blood chemistry tests and urinalysis, including urine sample for drug screening;
* A negative urine drug test (barbiturates, benzodiazepines, amphetamines, opiates, cocaine, cannabinoids, ethanol) at screening, and at each laboratory day;
* Subjects must be non-smokers. A breath sample analysis will be conducted on-site with an Alco-Sensor Intoximeter, and an Innovative Medical Monitoring carbon monoxide (CO) Monitor, and must reveal a CO value of less than or equal to 8 ppm and a negative cotinine urine or saliva test (>100 ng/mL);
* Females must have a negative pregnancy test (beta human chorionic gonadotrophin) at screening, and prior to each study drug administration. Females capable of childbearing are required to use a medically accepted form of contraception for at least 1 month prior to study start, throughout the study duration, and for at least 1 month after study medication is discontinued.

Exclusion Criteria:

* Current participation in the follow-up period of a preceding drug research study;
* Presence of unresolved/unstable psychiatric comorbidities as determined by clinical assessment and structured clinical interview using the SCID-1, that could interfere with study evaluations or affect a subject's safety;
* Recent history of drug addiction and/or alcoholism; and nicotine dependence within the past 6 months, as determined by psychiatric clinical assessment;
* Current significant acute or chronic medical disease, or any historical medical condition that could relapse during or immediately after the study and, in the investigator's opinion, may interfere with study evaluations or affect a subject's safety;
* Presence of potential organic etiology (e.g., a serious head injury or injury resulting in loss of consciousness, seizure disorder, thyroid problems, etc.) for ADHD symptomatology, as determined by clinical assessment;
* Blood pressure over 160/100 mmHg or under 90/40 mmHg, or heart rate over 120 beats per minute or below 40 beats per minute, obtained on two consecutive measures over 15 minutes when the subject is at rest;
* Exposure to any investigational new drug within 30 days of screening;
* Regular use of any prescription, over-the-counter drugs or likely need for concomitant treatment medication during the study period;
* Use of herbal products, including St. John's Wort, for 2 weeks prior to study initiation and throughout the study duration.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2008-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Attention as measured by Conners' Continuous Performance Task(CPT) | Measured at Lab Visits 1 through 7
Impulsivity as measured by the CPT and Stop Signal Reaction Test | Measured at Lab Visits 1 through 7
Working memory as measured by Digit Span Backwards and Two-Back Test | Measured at Lab Visits 1 through 7

SECONDARY OUTCOMES:
Subjective effects | Measured at Lab Visits 1 through 7
Cardiovascular effects | Measured at Lab Visits 1 through 7
Drug effects | Measured at Lab Visits 1 through 7

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A. Martin, MD, Principal Investigator — University of Kentucky Department of Psychiatry
Locations (1):
- General Clinical Research Center, University of Kentucky, Lexington, Kentucky, United States